CLINICAL TRIAL: NCT02834533
Title: Robotic Gait Training in Multiple Sclerosis: a Randomized Clinical Trial Evaluating Virtual Reality Role
Brief Title: Role of Virtual Reality in MS Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Prof, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/2014
Record Dates: First submitted 2016-07-04; First posted 2016-07-15 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis Relapse
Keywords: Lokomat;; robotic rehabilitation.; Multiple Sclerosis;; Virtual reality
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- column heading in tables. (Active Comparator): The group 1 (G1, n=20) underwent Lokomat-Nanos training. Each patient underwent 40 1h-training sessions (for 3 times a week). Both the study groups were treated by Lokomat (Hocoma Inc., Zurich, Switzerland), which includes a treadmill, a BWSS and two powered gait orthosis robotic actuators with integrated computer-controlled linear actuators at each hip and knee joint . The overall duration of Lokomat therapy, including the time to get on and off, was 60min, while the robotic gait training lasted around 40min.
  Interventions: Device: Lokomat
- row and column in table (Active Comparator): The group 2 (G2, n=20) underwent Lokomat-Pro training, with the same G1 sessions. The Pro device offers instead a VR through an Augmented Feedback Module, which provides instructive, stimulating, interactive, and direct feedbacks to enhance the patient's motivation by projecting his/her avatar while walking on a screen.
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — Lokomat (Hocoma Inc., Zurich, Switzerland)includes a treadmill, a BWSS and two powered gait orthosis robotic actuators with integrated computer-controlled linear actuators at each hip and knee joint . As compared to Lokomat-Nanos, the Pro device offers a VR through an Augmented Feedback Module, which provides instructive, stimulating, interactive, and direct feedbacks to enhance the patient's motivation by projecting his/her avatar while walking on a screen.

SUMMARY:
Objective: To investigate the role of virtual reality (VR) paired with robotic-assisted gait training (RAGT) compared with RAGT alone in patients with Multiple Sclerosis (MS).

Method: A Randomized, double-blind, controlled clinical trial was carried out in forty patients with relapsing remitting MS. All patients were randomized into two groups. One group practiced Lokomat without VR (group G1), the other one the Lokomat with VR (G2). Both the groups performed 40-1h-training sessions by Lokomat (for 3 times a week). A skilled-blinded neurologist and psychologist administered clinical and neuropsychological scales. All the clinical tests were performed at the beginning (T0) and at the end (T1) of the rehabilitative program.

DETAILED DESCRIPTION:
METHODS The present study is a single-blind randomized trial, conducted according to the Declaration of Helsinki, the guidelines for Good Clinical Practice, and the (CONSORT) Statement guidelines. The study protocol was approved by our Institutional Review Board and Ethics Committee (project number: 24/2013).

One hundred and fifty consecutive outpatients with relapsing-remitting multiple sclerosis and gait and/or balance disturbance, attending the Laboratory of Robotic Neurorehabilitation of the IRCCS Neurolesi Bonino-Pulejo (Messina, Italy) from January 2015 to January 2016, were invited to participate in the study, and were screened for study eligibility.

Inclusion/exclusion criteria Inclusion criteria were: age 30-65 years; severe walking disability with Expanded Disability Status Score between 3.5 and 6.0 (Piramidal subitem ≥3); Montreal Cognitive Assessment score ≥24; absence of concomitant neurological or orthopedic conditions that may interfere with ambulation; stable pharmacological therapy for at least 6 months. Exclusion criteria were: multiple sclerosis relapse during the three months prior to recruitment; presence of paroxysmal vertigo; lower limb botulinum toxin injections within the previous 12 weeks; cardiorespiratory instability; high-risk of spontaneous fracture; lower-limb skin lesions and phlebitis/thrombosis; more than 130 kg body weight.

Randomization Forty out of 150 outpatients with relapsing remitting multiple sclerosis form, according to Polman criteria14 selected between January 2015-2016, were enrolled and randomized and allocated into either Group1 (G1 i.e. Lokomat-Nanos) or Group2 (G2 i.e. Lokomat-Pro), as shown in fig 1. The subjects were randomly assigned to one of two treatment groups, using a simple randomization scheme generated by a software (www.randomization.com). Individual, sequentially numbered index cards with the random assignments were prepared. The index cards were folded and placed in sealed opaque envelopes. A physician member of the research team, who was blinded to the baseline examination findings, opened the envelopes to attribute the interventions according to the group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Severe walking disability with Expanded Disability Status Score (EDSS) between 3.5 and 6.0 (Pyramidal subitem ≥3)
* Montreal Cognitive Assessment score ≥24
* Absence of concomitant neurological or orthopedic conditions that may interfere with ambulation.

Exclusion Criteria:

* MS relapse during the three months prior to recruitment
* Not well defined pharmacological therapy; presence of paroxysmal vertigo
* Lower limb botulinum toxin injections within the previous 12 weeks
* Cardiorespiratory instability high-risk of spontaneous fracture
* Lower-limb skin lesions and phlebitis/thrombosis
* More than 130kg body weight

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Up to 14 weeks
  BBS is a clinical scale to evaluate balance

SECONDARY OUTCOMES:
Coping Orientation to Problem Experienced | Up to 14 weeks
  The test is aimed at evaluating how a person deals with a specific problem, with two main coping strategies, i.e. adaptation and avoidance.

IPD SHARING:
Plan to Share IPD: Undecided
We are planning this.